CLINICAL TRIAL: NCT02075528
Title: Early Prediction of Clinical Response, Metabolic Change, and Pharmacokinetics in Taiwanese Patients With Schizophrenia Patients Treated by Paliperidone ER: an Open-Label Study
Brief Title: Early Prediction of Clinical Response in Patients With Schizophrenia Treated by Paliperidone ER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: Johnson & Johnson Taiwan Ltd (Industry); Taipei Institute of Pathology (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPP-2009-OLS
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Paliperidone; Treatment response; Schizophrenia; Early prediction; Pharmacokinetics
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paliperidone Extended Release (ER) (Experimental): The participants were assigned to receive a fixed dosage of 9 mg/d of paliperidone ER for the first 2 weeks. The paliperidone ER dosage was adjusted flexibly after 2 weeks according to the clinical judgment of the physicians in charge.
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — 9 mg/d of paliperidone ER was administered during the first 2 weeks, after which the dose was adjusted clinically
  Other Names: 9-hydroxyrisperidone

SUMMARY:
Paliperidone ER is a new psychotropic medication for schizophrenia treatment. The studies of 6-week acute treatment and 52-week maintenance treatment showed positive results in patients with schizophrenia and its clinical improvement may start at Day 4. Some second-generation antipsychotics have been found that using the first 2 weeks' treatment results to predict the fourth or sixth week's treatment response is acceptable.

The primary aim of this study is to investigate:

1. . whether the early prediction model used in other atypicals could also be applied in paliperidone ER.
2. . The changes of metabolic parameters and pharmacokinetics after paliperidone ER treatment in this study

DETAILED DESCRIPTION:
Patients diagnosed with schizophrenia or schizoaffective disorders will be enrolled in the 6-week trial. Eligible patients will receive 9mg paliperidone ER first. Then, the dosage of paliperidone could be adjusted two weeks later according to clinical judgement. They will be followed and receive assessment of pharmacokinetics, metabolic parameters ( lipid profiles, glucose, insulin, adiponectin, leptin, and prolactin, etc.), and the treatment response.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* a minimal baseline total score of 60 on the PANSS
* those who had not received long-acting antipsychotic injection for the preceding 6 months
* physically healthy and standard clinical laboratory test results within laboratory reference ranges, or if outside the ranges, judged to be clinically insignificant by the investigators.

Exclusion Criteria:

* diagnosis of substance (including alcohol) dependence in the previous 6 months
* a medical condition that could affect absorption, metabolism, or excretion of the study drug
* substantial risk of suicide or violent behavior
* pregnancy or breastfeeding
* documented organic disease of the central nervous system
* unstable or critical untreated medical illness
* history of clozapine treatment in the previous 3 months
* participation in an investigational drug trial in the 30 days before screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Responder: more than 50% improvement on the total score of the Positive and Negative Syndrome Scale (PANSS) | Baseline (day 0) and Day 42

SECONDARY OUTCOMES:
Metabolic parameters(including lipid profiles, fasting glucose, adiponectin, leptin, and insulin, and prolactin) | Day 0 and 42

OTHER OUTCOMES:
pharmacokinetic (levels of 9-OH risperidone) | day 14 and day 42

CONTACTS AND LOCATIONS:
Overall Officials: MING-CHYI HUANG, M.D., Ph.D., Principal Investigator — Department of Psychiatry, Taipei City Hospital, Songde Branch, Taipei, Taiwan
Locations (1):
- Taipei City Hospital, Songde Branch, Taipei, Taiwan